CLINICAL TRIAL: NCT06177314
Title: Molecular Diagnosis of Allergic Contact Dermatitis
Acronym: MODAL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 23-5132; 69HCL23_1277 (Other: Eaysdore)
Record Dates: First submitted 2023-12-11; First posted 2023-12-20 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Contact Dermatitis; Contact Dermatitis Irritant; Contact Dermatitis, Allergic
Keywords: allergic contact dermatitis; irritant contact dermatitis; molecular signature; transcriptomic profiling; biomarkers; point of care diagnosis
MeSH Terms: conditions — Dermatitis, Contact; Dermatitis, Irritant; Dermatitis, Allergic Contact

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Active contact dermatitis: patient suffering from contact dermatitis and presenting active cllinical lesions. Allergic or non allergic form of contact dermatitis was diagnose based on patch-test results and exposure assessment
  Interventions: Other: correlate the molecular signatures of active lesions of contact dermatitis with allergological results

INTERVENTIONS:
Other: correlate the molecular signatures of active lesions of contact dermatitis with allergological results — Data will be collected retrospectively and prospectively from patients' medical records, and will include: clinical information (history, treatments, lifestyle, exposures, lesion location and appearance), patch-test results, histological analysis results, molecular analysis results.

SUMMARY:
Allergic contact dermatitis (ACD) is a common inflammatory skin disease, affecting approximately 15-20% of the general population in industrialized countries and ranking first among occupational diseases in many European countries.

ACD typically presents as a severe skin inflammation with redness, edema, oozing and crusting. It is characterized by a delayed type IV hypersensitivity response mediated by allergen-specific T cells in sensitized individuals.

Current diagnosis relies on clinical investigations by diagnostic patch testing with suspected allergenic chemicals. The patch test method aims at reproducing the eczematous lesions by applying occlusive patches containing the suspected allergens to the patient's healthy skin. This is a time consuming and costly process. It requires experienced medical staff to read the reaction, and is only performed by a limited number of expert dermato-allergologists across Europe (which limits the accessibility of suspected ACD patients to diagnosis). Finally, if the robustness of the patch-test method is undisputable, it cannot be neglected that patch-test results are sometimes false positive or non-relevant, which leads to non-appropriate disease management.

Therefore, there is today an urgent need for the availability of new ex vivo/in vitro tools based on the modern understanding of the immune mechanisms of ACD to enhance the current diagnostic procedure, and open new avenues for a personalized diagnosis of skin ACD.

In this context, the team "Epidermal Immunity and Allergy" (CIRI, Inserm U1111) recently characterized the molecular signatures of ACD (using microarrays), based on positive patch-test reactions to reference chemical allergens or non-allergenic irritants. It was shown that there are unique molecular profiles and signaling pathways characterizing each inflammation. Machine learning methods were then developed to identify and validate classification algorithms based on the expression levels of a minimum set of biomarkers (n=12), enabling very good discrimination between allergen-induced and irritant-induced patch-test inflammation (which was confirmed by complementary quantitative RT-PCR analyses). Finally, some patients with weak positive patch-test reactions to allergens show no/low marks of allergy molecular signature, questioning about the reliability/relevance of their patch-tests results.

Our results therefore stress the value of molecular profiling of patch-test reactions to improve/reinforce clinical ACD diagnosis, and to help the dermatologist to discriminate true versus false positive patch test reactions.

Importantly, those results also open new avenues for the development of a future point care diagnosis. Indeed, it is currently is estimated that only 20% of patients being sent for allergology work-ups suffer from true skin allergy (i.e. patients with positive patch-tests, combined with relevant clinical history and confirmatory use tests). Most of the patients (80%) are in fact suffering from skin irritation. Therefore, the detection of ACD biomarkers in active eczema lesions could provide the dermatologist with major information to improve and accelerate its clinical diagnosis. This could also prevent numerous patients (negative for ACD biomarkers) being sent for unnecessary allergology work-ups.

However, to date, it remains to be demonstrated that (i) the same panel of ACD biomarkers is expressed both in acute eczema lesions and positive patch-test reactions, and that (ii) the detection of these biomarkers allows for a sensitive and reliable diagnosis of skin allergy.

The main objective of the study will be to make the proof of concept that the expression of allergy biomarkers correlates with patients suffering from true ACD (i.e. patients with high biomarker expression in acute lesions, positive patch-tests and relevant clinical history), versus those developing skin irritation (no/low biomarker expression in acute lesions, negative patch-tests, and lack of clinical history).

ELIGIBILITY:
Inclusion Criteria:

* Patient, male or female, over 18 years of age
* Patient with active contact dermatitis lesion biopsied for molecular analysis
* Patients who have undergone patch testing
* Patients whose positive patch tests were biopsied for molecular analysis
* Written informed consent given prior to any study-related procedure
* Between 01/01/2020 and 31/12/2025

Exclusion Criteria:

* Missing clinical data
* Patient objecting to use of data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred for suspected contact dermatitis to the Allergology and Clinical Immunology Department of the Centre Hospitalier Lyon Sud and the Dermatology and Allergology Department of the Centre Hospitalier Universitaire de St Etienne, with active eczema lesions, and who benefited from skin biopsies and allergoly work-up (patch tests) as part of their management.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
expression levels of allergy biomarkers | during standard of care
  expression levels of allergy biomarkers, expressed as fold change (ratio between gene expression levels in lesional skin of active dermatitis lesions and their expression levels in healthy skin of the same patient)

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Lyon Sud, Pierre-Bénite, France